CLINICAL TRIAL: NCT02546713
Title: The Influence of Abutment Macro-design on Peri-implant Tissue Dimensions for Guided Placed and Restored Implants
Brief Title: Abutment Macro Design and Peri-implant Tissues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Collaborators: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Principal Investigator, Theofilos Koutouzis, Associate Professor, Nova Southeastern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: I-AA-14-075
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Edentulous
Keywords: dental implants
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Other): Abutments with a concave configuration of the subcritical contour (emergence shape).
  Interventions: Other: Abutment with concave subcritical contour
- Group 2 (Other): Abutments with convex configuration of the subcritical contour (emergence shape)
  Interventions: Other: Abutment with convex subcritical contour

INTERVENTIONS:
Other: Abutment with concave subcritical contour — Implants will be restored with abutments with concave configuration of the subcritical contour
  Arms: Group 1
Other: Abutment with convex subcritical contour — Implants will be restored with abutments with convex configuration of the subcritical contour
  Arms: Group 2

SUMMARY:
The aim of this study is to evaluate the effect of abutment macro-design on soft and hard tissue responses. This trial is designed as a randomized controlled clinical study in which two groups of fourteen partially edentulous patients will have as part of their treatment one implant placed in the maxillary premolar region.

DETAILED DESCRIPTION:
Implant placement and abutment design will be planned with a computer software for guided implant treatment (SIMPLANT). The surgical implant placement will be performed under manufacturer's protocol by placing the implant platform 1mm below the buccal aspect of the osteotomy (Koutouzis et al 2013). Virtually designed, permanent CAD-CAM fabricated abutments (ATLANTIS, DENTSPLY) with different configuration of the subcritical contour (emergence shape) will be connected to the implants and temporary crowns will be delivered.

Implants of the Group 1 will have permanent abutments with a concave configuration of the subcritical contour (emergence shape).

Implants of the Group 2 will have permanent abutments with a convex configuration of the subcritical contour (emergence shape).

The patients will be restored with single crowns 3 months following implant installation.

A randomization protocol will be produced from a computer-generated list for the distribution of subjects in the two treatment groups.

ELIGIBILITY:
General Inclusion criteria:

* - Age more than 21 years
* Absence of relevant medical conditions
* Availability for 12 month follow-up

Specific Inclusion criteria:

* One missing tooth in the maxillary premolar region
* Presence of two adjacent teeth at the implant site
* Absence of periodontal disease
* Healed osseous architecture enough to receive an implant with a diameter of at least 3.5 mm and a sufficient amount of bone for placing implants with a length of at least 9 mm

General Exclusion Criteria:

* - Pregnancy at the screening visit.
* Smoking more than 10 cig/day

Specific Exclusion criteria:

* Adjacent implants
* Presence of periapical radiolucency at the adjacent teeth
* Missing adjacent teeth

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Peri-implant mucosa margin position change | Day 7-10 to the Day 360
  The primary outcome variable will be change on peri-implant mucosa margin position.

CONTACTS AND LOCATIONS:
Overall Officials: Theofilos Koutouzis, DDS, Principal Investigator — Nova Southeastern University
Locations (1):
- Nova Southeastern University, Fort Lauderdale, Florida, United States

REFERENCES:
- [Background] Koutouzis T, Neiva R, Nair M, Nonhoff J, Lundgren T. Cone beam computed tomographic evaluation of implants with platform-switched Morse taper connection with the implant-abutment interface at different levels in relation to the alveolar crest. Int J Oral Maxillofac Implants. 2014 Sep-Oct;29(5):1157-63. doi: 10.11607/jomi.3411. PMID 25216143
- [Background] Koutouzis T, Koutouzis G, Tomasi C, Lundgren T. Immediate loading of implants placed with the osteotome technique: one-year prospective case series. J Periodontol. 2011 Nov;82(11):1556-62. doi: 10.1902/jop.2011.100751. Epub 2011 May 4. PMID 21542730